CLINICAL TRIAL: NCT00122278
Title: Parenteral Corticosteroids as Adjuvant Therapy for Migraine Headaches
Brief Title: Headache in the Emergency Department (ED) - A Multi-Center Research Network to Optimize the ED Treatment of Migraines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Benjamin W. Friedman, MD, Prof. Emergency Medicine, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 05-02-032S
Record Dates: First submitted 2005-07-20; First posted 2005-07-22 (Estimated); Results first posted 2018-11-13 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-04

CONDITIONS: Migraine
Keywords: migraine, emergency department, dexamethasone; Migraine with or without aura or probable migraine without aura as defined by ICHD, 2nd edition
MeSH Terms: conditions — Migraine Disorders; Emergencies | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes

ARMS (2):
- Dexamethasone (Experimental): Dexamethasone 10 mg
  Interventions: Drug: Dexamethasone
- Placebo (Placebo Comparator): Placebo Dexamethasone, 10 mg
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone 10mg IV
  Other Names: Parental corticosteroid
  Arms: Dexamethasone
Other: Placebo — Placebo Dexamethasone 10mg IV
  Arms: Placebo

SUMMARY:
Migraines are a specific type of headache that frequently recur and are very painful. Although there are many medications that are effective against migraines, none of these medications cure 100% of migraines. Another problem with migraines is that although many times they get better after intravenous (IV) treatment in the emergency room (ER), about 1/3 of the time migraines recur the next day. The purpose of this research project is to see if adding a medication called dexamethasone to standard ER therapy will help patients get better quicker and stay pain-free more often than if they receive placebo.

DETAILED DESCRIPTION:
Parenteral Corticosteroids as Adjuvant Therapy for Migraine Headaches:

A. Overview/Aims: Five million Americans present to emergency departments (ED) annually with headaches [1]. The majority of these patients have migraine headaches [2,3]. Parenteral medications of proven benefit for acute migraines include the triptans [4], dopamine-receptor antagonists [5-11], non-steroidals [12], and dihydroergotamine [13]. Although these distinct classes of medication are often effective for the treatment of acute migraines, their use is complicated by treatment failures [4,9,14], recurrence of headache [15,16], and side effects [17], all of which are of concern for patients with migraines [18]. The ideal medication, which would rapidly alleviate migraine pain without any recurrence of pain or side effects, has not yet been identified.

The role of corticosteroids in acute migraines is ill-defined. Although used in patients with intractable migraines, this class of medication is not widely used in typical migraine attacks. However, limited clinical data suggest that corticosteroids decrease the rate of recurrent headaches [19-21] and might decrease the pain of an acute attack [22]. Further research is needed to define the role of corticosteroids in the ED treatment of acute migraine headaches.

Specific Aim: The specific aim of this study is to determine the efficacy of ten milligrams of parenteral dexamethasone as adjuvant therapy for the emergency department treatment of migraine headaches.

Primary Hypothesis: Twenty four hours after medication administration, a greater percentage of migraine subjects who received dexamethasone will have:

* sustained pain-free headache relief; and
* no headache-related functional impairment when compared to subjects who receive placebo.

Both groups will also receive the standard of care.

Secondary Hypothesis: Two hours after medication administration, a greater percentage of migraine subjects who received dexamethasone will be headache pain-free, when compared to subjects who receive placebo.

B. Background and Significance:

Despite standard treatment, a large percentage of emergency migraineurs continue to suffer from headaches after ED discharge. Recurrent or persistent headaches rated as moderate or severe in intensity occurred in 14-43% of subjects 24 hours after discharge in ED-based migraine clinical trials [20,23,24]. In a Canadian population, 45% of headache patients reported headache-related functional impairment within 24 hours of ED discharge [16].

Some reports indicate that corticosteroids decrease the rate and intensity of recurrent migraine headaches [19-21]. However, the investigators could not find any corticosteroid clinical trials using recommended measures and outcomes [25] in a migraine population. To the best of their knowledge, no controlled clinical trial has tested the efficacy of corticosteroids as primary migraine-abortive therapy.

Although the pathogenesis of migraine headaches is incompletely understood, a sterile neurogenic inflammation is felt to be key to the pain generating pathway that occurs in acute migraines [15]. Corticosteroids theoretically mitigate this inflammation and decrease the pain and duration of acute migraine attacks.

One dose of intravenous dexamethasone has been well-tolerated in migraineurs [20]. If this medication proves to have efficacy for migraines, then this would represent a substantial contribution to headache medicine, an effective tool in the armamentarium of emergency physicians, and a cheap and safe method to decrease the pain and suffering of ED migraine patients.

C. Methods:

C1. Overview: This will be a randomized, double-blind, placebo-controlled clinical research trial testing the efficacy of intravenous dexamethasone sodium phosphate as adjuvant therapy for acute migraine headaches. All subjects will receive standard-of-care migraine-abortive medication for their migraines. In addition, they will receive either ten milligrams of intravenous dexamethasone sodium phosphate or a comparable amount of placebo. Subjects will be followed by telephone 24 hours after medication administration.

C2. Study Sites: Study sites will include the emergency departments of Montefiore Medical Center, Jacobi Medical Center, New York Presbyterian Hospital, St. Luke's Medical Center, Bellevue Medical Center, and Kings County Medical Center.

C3. Selection of Participants: The attending emergency physician will refer all adult patients who present with a chief complaint of headache during the regular hours of the data collectors. Under the supervision of the site investigators, the data collectors will inform patients about the study and ask for their consent to participate in this study as human subjects. The data collectors will include in this study any patient who has a migraine headache as defined by the International Headache Society (IHS-2003 1.1 migraine without aura; 1.2 migraine with aura). Patients will also be included if they have an IHS probable migraine (IHS-2003 1.6.1 & 1.6.2) [26] that has lasted between 72 and 168 hours. In other words, patients will also be included if their headache meets all IHS migraine criteria except that the duration of the headache has been between 73 and 168 hours. These probable migraine patients will be included because they represent a substantial subset of ED primary headache patients (Friedman, et. al., unpublished data) and because the majority of patients with a disabling probable migraine and a history of similar headaches will respond to migraine-specific medication [27].

Patients will be excluded if the emergency physician intends to perform a lumbar puncture in the ED because lumbar puncture has an independent association with 24 hour headache pain scores. Patients will be excluded for persistent objective focal neurologic deficits, as determined by the attending physician, for fear of mistaking a stroke for a complicated migraine, or for signs and symptoms concerning for other causes of malignant secondary headache such as meningitis, subarachnoid hemorrhage, carotid dissection, or intracranial mass. Patients will also be excluded for temperatures greater than 100.3 degrees, pregnancy or lactation, or allergy or intolerance to any of the study medications. Patients can only enroll once. Patients over the age of 64 will be excluded, for fear of increased risk of adverse reactions to study medications and increased risk of secondary headaches. Patients who do not meet enrollment criteria will have basic demographic and headache variables recorded.

C4. Randomization and Blinding: Randomization is to be done by the research pharmacist at Montefiore Medical Center in blocks of six using computer generated random number tables available online. The randomization will be stratified by study site. In an order determined by the random number tables, the pharmacist will insert medication into vials and place these vials into sequentially numbered brown paper research bags. The research bags will be distributed by express courier in batches of six to the investigators at each site. The research bags will be stored at each site in a locked location accessible to the data collectors. When a subject has been identified, the contents of each research bag will be administered by a clinical nurse. Assignment will be known only by the research pharmacist. However, the assignment will accompany each research bag, sealed in a small manila envelope, in case a medical emergency mandates that the assignment be revealed.

C5. Measures:

C5a. Categorical Scale: As a primary measure, this trial will use the four point descriptive scale recommended for use in migraine research [25]. On this scale, subjects are asked to characterize their migraine pain as "none, mild, moderate or severe".

C5b. Disability Scale: A descriptive categorical scale will be used to characterize the subject's headache-related disability. On this scale, subjects describe their disability as "1) none; 2) mildly impaired (having a little bit of difficulty doing what I usually do); 3) moderately impaired (having a great deal of difficulty doing what I usually do and can only do very minor activities); or 4) severely impaired (requiring bed rest)" [25].

C5c. Numerical Rating Scale for Pain: An 11-point verbal numerical rating scale for pain will be a secondary measurement tool for this trial. On this scale, subjects are asked to describe their pain as a number between zero and ten, with zero being no pain and ten being the worst pain imaginable. This scale has been shown to perform comparably to a visual analog scale, while being easier to administer [28].

C6.Outcomes: The primary outcome will be the percentage of subjects who achieve and maintain a "headache pain free" state. Persistent "headache pain free" is the recommended outcome for migraine clinical research [25]. Subjects will be considered to have fulfilled the primary outcome if they achieve a pain free state in the ED and maintain this throughout the 24 hour period after receiving study medication. The alternate primary outcome will be the number of subjects who report no headache-related disability for the period of time after ED discharge. The major secondary outcome will be the percentage of subjects who report a "headache pain-free" status two hours after medication administration.

Other secondary outcomes include rates of sustained headache relief (moderate or severe pain becoming and maintaining a level of mild or none), two-hour NRS change (NRSbaseline-NRS2hours), 24 hour NRS change (NRSbaseline-NRS24hours), need for rescue medication before two hours, need for analgesic medication after discharge from the ED, associated symptoms (specifically: weakness, drowsiness, dizziness), unscheduled visits to a medical provider within 24 hours of medication administration, and the percentage of patients who answer affirmatively to the question "Do you want to receive the same medication the next time you come to the ED?"

C7. Data Collection, Data Entry, and Back-Up: Data entry and follow-up of subjects will be accomplished by taking advantage of the research infrastructure in place at the Department of Emergency Medicine of the Albert Einstein College of Medicine. Five full-time research assistants and one research clerk are funded by the department. The research assistants are medical technician level, full-time employees who have extensive clinical research experience and have passed required research ethics courses. These research assistants staff the Montefiore ED during all operational hours.

The initial data collection process will be performed by the data collectors at each individual site. These data collectors will be different in each ED, depending on the resources at the individual ED. At Montefiore and Jacobi, the data collectors are salaried, trained, technician level employees, who have passed required research ethics courses. The data collectors will be trained for this particular study by the principal investigator and site investigators. Their training will include mock patient encounters. The data collectors will use a standardized data collection instrument to collect baseline information, pain scores, and side effects in the ED. After the ED data have been obtained, the data collection instrument will be photocopied and faxed to a dedicated research clerk in the Department of Emergency Medicine at Albert Einstein College of Medicine. The receiving fax machine is a private fax machine secured in an office behind two locked doors.

The research clerk will be responsible for obtaining the 24 hour follow-up information. At a time pre-arranged with the subject prior to the subject's discharge from the ED, the research clerk will call the subject and obtain 24 hour follow-up information by reading questions off of the data collection instrument. Twenty-four hour follow-up to be done during non-business hours will be performed by Montefiore's research assistants, who cover the ED 24 hours a day, seven days every week. These research assistants will retrieve the faxed data collection instruments, obtain the follow-up information, and then return the data collection instruments to the research clerk.

The research clerk will enter all data into SPSS data entry V.11. Completed data collection instruments will be sent to a second research clerk who will enter the data a second time into the same SPSS program. After every ten subjects have been entered, data will be backed up and stored on three different computers on two distinct campuses. Prior to all analyses, the two data sets will be compared. Discrepancies will be corrected using the initial data collection instrument as the source. The original version of each data collection instrument will be kept in a locked cabinet at its original site.

C8. Medications: In addition to study medication or placebo, all subjects will receive standard migraine abortive therapy. The optimal migraine-abortive/analgesic medication for ED patients with acute migraine headaches has not yet been defined, so the investigators have chosen intravenous metoclopramide, an effective, safe, widely-available, and economical dopamine receptor antagonist, as the migraine treatment for this trial. Parenteral dopamine-antagonists are recommended for use in the ED29 and are used more commonly than triptans in the ED setting [1,16]. Metoclopramide has been shown to be at least as effective as subcutaneous sumatriptan at reducing pain [7,8] with comparable two hour activity limitations [30]. The investigators will use 20 milligrams of intravenous metoclopramide, a moderate dose when compared to their previous work [23,30]. In addition to metoclopramide, each subject will also receive 25mg of diphenhydramine to prevent akathisia and other extra-pyramidal reactions to the metoclopramide [31]. This combination of metoclopramide and diphenhydramine is commonly used in the ED setting and does not cause significant drowsiness or impairment of activities in migraineurs at two hours [30]. The investigators view the potential anti-migraine effect of diphenhydramine [32] as added benefit for their subjects. Metoclopramide, diphenhydramine, and the study medication will be placed into a 50cc bag of normal saline and administered as a slow intravenous drip over twenty minutes.

Subjects who require rescue medication for persistent headache will receive another 20mg of intravenous metoclopramide. This additional dose of metoclopramide is part of an ED-based protocol that has demonstrated a high rate of pain relief and patient satisfaction with a minimum of side effects [23,30].

Subjects who require more pain medication will receive a combination of ibuprofen and oral opiates at the discretion of the treating physician.

All subjects will be discharged from the ED with two 400mg tablets of ibuprofen to be taken as needed for recurrence of headache. Ibuprofen is an effective migraine treatment [9].

C9. Interim Analysis, Stopping Rules and Sample Size Calculation: An interim analysis will be performed to detect an overwhelming superiority of the intervention. A data monitoring committee will convene after 126 subjects have been enrolled. The committee will look for a statistically significant difference in the primary outcome or a discrepancy in the rate of adverse effects (measured by rate of hospitalization for presumed adverse reaction to medication). The medications used in this study are well-known to the medical community and commonly used. Neither the disease nor the medications cause mortality or significant permanent disability. Therefore, although the investigators will monitor the adverse effects that occur during this trial, they do not anticipate that this will have a significant effect on the outcome.

There are many different approaches to calculation of significance criteria that can be used in interim analyses, and thus might be used to terminate a trial before the complete data are collected. The investigators have chosen an intermediate approach, based on the O'Brien-Fleming procedure [33] and set the interim test criterion at 0.01, and the final test criterion at 0.04. Using a criterion for significance of 0.04 and a 2-tailed test, this study will require 100 subjects in each group, for a total of 200 subjects, to have power of 80% to yield a statistically significant result. This computation assumes that the difference in persistent headache pain-free proportions is 0.20, specifically, 0.30 versus 0.50 (the rate of persistent headache pain-free 24 hours after ED discharge in a previous similarly-dosed metoclopramide trial was 30% [30]). The clinical effect being sought is comparable to a number needed to treat of five, the largest number needed to treat believed important to discover for this self-limited disease process. The interim analysis will have adequate power (0.80) to discover a statistically significant difference (alpha=0.01) if the difference between the two groups is 30% (.60 versus .30).

C10. Co-Variates: The following variables will be assessed:

C10a. Cutaneous Allodynia: Cutaneous allodynia is felt to be a marker of more intractable migraines [34] and can be tested for by lightly rubbing a 4 x 4 piece of gauze on the face of the subject [35]. The data collectors will assess each subject for cutaneous allodynia prior to the administration of medication.

C10b. Duration of Headache: Although likely to be collinear with allodynia, this co-variate might be associated with intractable 24 hour headaches [20].

C10c. Pre-Medication: In previous work, although 25% of the investigators' population took no analgesic medication prior to presentation to the ED, this co-variate did not confound the association between study medication and persistent pain-free [30]. Nevertheless, the investigators will record all migraine-relevant medications used by their subjects prior to ED presentation, group these by class, and determine if this co-variate has a relationship with the primary outcomes.

C11d. Aura: The investigators know of no documented association between aura and corticosteroids, but this subject has been inadequately explored.

C11e. Prophylactic Medications: In previous work [30], only a small minority of ED migraineurs were on prophylactic medication. However, these patients represent a sub-set of migraineurs with more severe disease.

C11f. Chronic Migraines: Only a small minority of ED migraineurs can be classified as chronic (Friedman, unpublished data). However, these patients represent a sub-set of migraineurs at high risk of recurrent 24 hour headaches.

C11g. Medication-Rebound Headaches: This diagnosis has been inadequately explored in the ED setting and consists of complicated headache patients. The investigators will not exclude these patients from this study because they are likely to benefit from this intervention [21].

C11h. Site: To account for site-specific differences from influencing the results, subjects from each site will be randomized in blocks of six to prevent unequal representation of a particular site in either arm. This will prevent any one site from overly influencing the study.

C11i. Race/Ethnicity: This will be based on subject's report. The significance of this co-variate for this study is unknown.

C11j. Age: This will be recorded. The significance of this co-variate for this study is unknown.

C12k.Gender: This will be recorded. The significance of this co-variate for this study is unknown.

C12. Analysis: The data will be analyzed in an "intention-to-treat" manner. Once a patient is randomized and receives the dexamethasone, their pain scores will be included in the 24-hour analysis regardless of whether or not they received rescue medication or completed the protocol. However, lost-to-follow-up subjects will be excluded from the primary analysis (a sensitivity analysis will be conducted in which lost-to-follow-up subjects are assumed to have a poor outcome). Study enrollment will continue until the pre-determined number of subjects have completed the primary endpoint. Chi-square analysis will be used to compare rates. Students t-tests will be used to compare mean differences in pain scores. Multivariate regression models will be used to analyze the influence of the co-variates discussed above, particularly allodynia, duration of headache, and use of medication prior to ED presentation. Briefly, evidence of confounding will be sought by looking for an association between the heterogeneous variable and both the independent (study medication) and dependent (pain status) variables. Between-group differences will be expressed as means or proportions, bounded by 95% confidence intervals (95% CI).

References:

1. Vinson DR. Treatment patterns of isolated benign headache in US emergency departments. Ann Emerg Med 2002; 39:215-22.
2. Bigal M, Bordini CA, Speciali JG. Headache in an emergency room in Brazil. Sao Paulo Med J 2000; 118:58-62.
3. Luda E, Comitangelo R, Sicuro L. The symptom of headache in emergency departments. The experience of a neurology emergency department. Ital J Neurol Sci 1995; 16:295-301.
4. Akpunonu BE, Mutgi AB, Federman DJ, et al. Subcutaneous sumatriptan for treatment of acute migraine in patients admitted to the emergency department: a multicenter study. Ann Emerg Med 1995; 25:464-9.
5. Bigal ME, Bordini CA, Speciali JG. Intravenous chlorpromazine in the emergency department treatment of migraines: a randomized controlled trial. J Emerg Med 2002; 23:141-8.
6. Kelly AM, Ardagh M, Curry C, D'Antonio J, Zebic S. Intravenous chlorpromazine versus intramuscular sumatriptan for acute migraine. J Accid Emerg Med 1997; 14:209-11.
7. Friedman B, Corbo J, Lipton R, et al. Metoclopramide Versus Sumatriptan for the ED Treatment of Migraines. Neurology 2005.
8. Esteban-Morales A, Chavez PT, Martinez CGR, Zuniga AS. Respuesta clinica de metoclopramida en comparacion con sumatriptan en el tratamiento de ataques agudos de migrana. Revista de la Sanidad Militar Mexico 1999; 53:36-40.
9. Tek DS, McClellan DS, Olshaker JS, Allen CL, Arthur DC. A prospective, double-blind study of metoclopramide hydrochloride for the control of migraine in the emergency department. Ann Emerg Med 1990; 19:1083-7.
10. Silberstein SD, Young WB, Mendizabal JE, Rothrock JF, Alam AS. Acute migraine treatment with droperidol: A randomized, double-blind, placebo-controlled trial. Neurology 2003; 60:315-21.
11. Seim MB, March JA, Dunn KA. Intravenous ketorolac vs intravenous prochlorperazine for the treatment of migraine headaches. Acad Emerg Med 1998; 5:573-6.
12. Meredith JT, Wait S, Brewer KL. A prospective double-blind study of nasal sumatriptan versus IV ketorolac in migraine. Am J Emerg Med 2003; 21:173-5.
13. Winner P, Ricalde O, Le Force B, Saper J, Margul B. A double-blind study of subcutaneous dihydroergotamine vs subcutaneous sumatriptan in the treatment of acute migraine. Arch Neurol 1996; 53:180-4.
14. Ellis GL, Delaney J, DeHart DA, Owens A. The efficacy of metoclopramide in the treatment of migraine headache. Ann Emerg Med 1993; 22:191-5.
15. Goadsby PJ, Lipton RB, Ferrari MD. Migraine--current understanding and treatment. N Engl J Med 2002; 346:257-70.
16. Ducharme J, Beveridge RC, Lee JS, Beaulieu S. Emergency management of migraine: is the headache really over? Acad Emerg Med 1998; 5:899-905.
17. Hardman J, Limbird L. Goodman and Gilman's the pharmacological basis of therapeutics, 9th ed. New York: McGraw-Hill, Health Professions Division, 1996.
18. Lipton RB, Hamelsky SW, Dayno JM. What do patients with migraine want from acute migraine treatment? Headache 2002; 42 Suppl 1:3-9.
19. Krymchantowski AV, Barbosa JS. Dexamethasone decreases migraine recurrence observed after treatment with a triptan combined with a nonsteroidal anti-inflammatory drug. Arq Neuropsiquiatr 2001; 59:708-11.
20. Innes G, Macphail I, Dillon E. Dexamethasone prevents relapse after emergency department treatment of acute migraine: a randomized clinical trial. Canadian Journal of Emergency Medicine 1999; 1.
21. Gallagher RM. Emergency treatment of intractable migraine. Headache 1986; 26:74-5.
22. Monzillo P, Nemoto P, Costa A, Sanvito W. Tratamento Agudo Da Crise De Enxaqueca Refrataria Na Emergencia. Arq Neuropsiquiatr 2004; 62:513-518.
23. Corbo J, Esses D, Bijur PE, Iannaccone R, Gallagher EJ. Randomized clinical trial of intravenous magnesium sulfate as an adjunctive medication for emergency department treatment of migraine headache. Ann Emerg Med 2001; 38:621-7.
24. Cameron JD, Lane PL, Speechley M. Intravenous chlorpromazine vs intravenous metoclopramide in acute migraine headache. Acad Emerg Med 1995; 2:597-602.
25. Tfelt-Hansen P, Block G, Dahlof C, et al. Guidelines for controlled trials of drugs in migraine: second edition. Cephalalgia 2000; 20:765-86.
26. Classification and diagnostic criteria for headache disorders, cranial neuralgias and facial pain. Headache Classification Committee of the International Headache Society. Cephalalgia 1988; 8 Suppl 7:1-96.
27. Lipton RB, Cady RK, Stewart WF, Wilks K, Hall C. Diagnostic lessons from the spectrum study. Neurology 2002; 58:S27-31.
28. Bijur PE, Latimer CT, Gallagher EJ. Validation of a verbally administered numerical rating scale of acute pain for use in the emergency department. Acad Emerg Med 2003; 10:390-2.
29. Kelly AM. Migraine: pharmacotherapy in the emergency department. J Accid Emerg Med 2000; 17:241-5.
30. Friedman BW, Corbo J, Lipton RB, et al. A trial of metoclopramide vs sumatriptan for the emergency department treatment of migraines. Neurology 2005; 64:463-8.
31. Drug Consult. St. Louis: Mosby, Inc., 2005.
32. Swidan SZ, Lake AE, 3rd, Saper JR. Efficacy of intravenous diphenhydramine versus intravenous DHE-45 in the treatment of severe migraine headache. Curr Pain Headache Rep 2005; 9:65-70.
33. O'Brien PC, Fleming TR. A multiple testing procedure for clinical trials. Biometrics 1979; 35:549-56.
34. Burstein R, Collins B, Jakubowski M. Defeating migraine pain with triptans: a race against the development of cutaneous allodynia. Ann Neurol 2004; 55:19-26.
35. Ashkenazi A, Sholtzow M, Young WB. Prevalence of Dynamic Mechanical (Brush) Allodynia in MIgraine (Abstract). Neurology 2004; 62:A83.

ELIGIBILITY:
Inclusion Criteria:

* Migraine with or without aura; probable migraine without aura

Exclusion Criteria:

* Secondary headache
* Allergy, contraindication or intolerance to study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2005-07; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin W. Friedman, MD, MS, Principal Investigator — Albert Einstein College of Medicine
Locations (3):
- United States (3):
  - Columbia University Medical Center, Manhattan, New York
  - St. Lukes Hospital, New York, New York
  - Jacobi Medical Center, The Bronx, New York

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexamethasone | Placebo
Started | 106 | 99
Completed | 104 | 99
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone | Placebo | Total
Number analyzed (Participants) | 106 | 99 | 205
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (10) | 37 (11) | 37 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 87 | 174
  Male | 19 | 12 | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 106 | 99 | 205
Duration of headache Prior to Study [Median (Inter-Quartile Range); unit: hours] | 48 [19 to 72] | 48 [12 to 72] | 48 [12 to 72]

OUTCOME MEASURES:

1. Primary Outcome: Persistent Headache Pain Free at 24 Hours
Description: Achieve headache freedom within two hours in the emergency department and no recurrence of pain within 24 hours of emergency department discharge
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 104 | 99
Participants | 26 | 19

2. Secondary Outcome: Functional Disability at 24 Hours
Description: No functional impairment within 24 hours of emergency department discharge
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 104 | 99
Participants | 70 | 55

ADVERSE EVENTS:
Arm/Group | Dexamethasone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/106 | 0/99
Serious Adverse Events (participants affected / at risk) | 0/106 | 0/99
Other Adverse Events (participants affected / at risk) | 41/106 | 27/99
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexamethasone (N=106) | Placebo (N=99)
Drowsiness (Nervous system disorders) | 19 (19) | 11 (11)
Dizziness (General disorders) | 3 (3) | 2 (2)
Acute Medication Reactoin (General disorders) | 10 (10) | 2 (2)
Other (General disorders) | 9 (9) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes